CLINICAL TRIAL: NCT00999115
Title: Clinical Trial in Phase I-IIa to Study the Feasibility and Security of the Allogenic Use of Adipose-derived Stem Cells for the Local Treatment of Recto-vaginal Fistula in Crohn´s Disease
Brief Title: Allogenic Stem Cells Derived From Lipoaspirates for the Treatment of Recto-vaginal Fistulas Associated to Crohn's Disease (ALOREVA)
Acronym: ALOREVA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Responsible Party: Principal Investigator, Ignacio Galicia, Professor, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC08/00153; EudraCT: 2009-010225-39
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Rectovaginal Fistula; Crohn Disease
Keywords: Rectovaginal Fistula; Crohn Disease; Allogenic; Adipose-Derived Stem Cells
MeSH Terms: conditions — Rectovaginal Fistula; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allogenic ASCs (Experimental): Intralesional dose of 20 million cells at baseline with a possible second administration of 40 million in case of incomplete fistula closure following week 12 assessment.
  Interventions: Drug: Expanded allogenic adipose-derived adult stem cells

INTERVENTIONS:
Drug: Expanded allogenic adipose-derived adult stem cells — Administration will be preceded by localization and closure of the internal opening. Cell treatment injection will be performed following Major Ambulatory Surgery standards. Patients will receive an intralesional dose of 20 million cells at baseline. 50% of the cell suspension will be placed into fistula walls of the internal opening, with the remaining 50% being injected across the wall tracts of the target fistula. Patients without healing (complete fistula closure)at week 12 will receive a second dose of 40 million cells, using the same treatment approach.
  Other Names: CX601 (company code)

SUMMARY:
The purpose of this study is to determine safety and efficacy of allogenic eASCs (expanded adult stem cells) for the treatment of recto-vaginal fistula in patients with Crohn´s disease.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patients with Crohn´s disease diagnosed at least 12 months earlier in accordance with accepted clinical, endoscopic, anatomopathological and/or radiologic criteria.
* Fulfilling one of the following criteria:

  * At least, one previous surgery for fistulous disease.
  * Physical status which discourage liposuction.
* Rectovaginal fistula.
* Women of a childbearing age. Good general state of health according to the findings of the clinical history and the physical examination.

Exclusion Criteria:

* Presence of severe proctitis (prominent friability, spontaneous bleeding, multiple erosions, deep ulcers) or dominant active luminal disease requiring immediate therapy, assessed by rectosigmoidoscopy
* Patients with CDAI≥201
* Patients with an abscess unless a complete toilet of the area with drainage of the collections and the absence of abscess and other collections is confirmed prior to treatment start
* Patients who have received infliximab or any other anti TNF agent in the 8 weeks before the cell treatment administration
* Patients who have received tacrolimus or cyclosporine in the 4 weeks before the cell treatment administration
* Patients with a history of abuse of alcohol or other addictive substances in the 6 months prior to inclusion
* Patients with malignant tumor, except for basal cell or cutaneous squamous cell carcinoma, or patients with a prior history of malignant tumors, unless the neoplastic disease has been in remission for the previous 5 years
* Patients with cardiopulmonary disease which, in opinion of the investigator, in unstable or sufficiently serious to exclude the patient from the study.
* Patients with any type of medical or psychiatric disease which, in the opinion of the investigator, could be grounds for exclusion from study
* Patients with congenital or acquired immunodeficiencies. HIV, HBV, HCV or treponema infection, whether active or latent.
* Patients allergic to local anesthetics or gadolinium (MRI contrast) MRI is unfeasible (e.g. due to the presence of pacemakers, hip replacements or severe claustrophobia)
* Patients who have suffering major surgery or severe trauma in the prior 6 months
* Pregnant or breastfeeding women
* Patients currently receiving, or having received within 1 month prior to enrolment into this clinical trial, any investigational drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in whom the external openings of the treated rectovaginal fistula have closed | 12 weeks

SECONDARY OUTCOMES:
Quality of life assessment using the SF-36 questionnaire | 12 weeks
Adverse events | 1, 4, 8,12, 24, 54 weeks
Clinically relevant variations in laboratory test | 1, 4 8, 12, 24, 54 weeks
Quality of life assessment using the SF-36 questionnaire | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Damián García Olmo, MD, Principal Investigator — General Surgery Department, Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Background] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Background] Garcia-Olmo D, Herreros D, Pascual M, Pascual I, De-La-Quintana P, Trebol J, Garcia-Arranz M. Treatment of enterocutaneous fistula in Crohn's Disease with adipose-derived stem cells: a comparison of protocols with and without cell expansion. Int J Colorectal Dis. 2009 Jan;24(1):27-30. doi: 10.1007/s00384-008-0559-0. Epub 2008 Aug 12. PMID 18696086
- [Background] Garcia-Olmo D, Garcia-Arranz M, Herreros D. Expanded adipose-derived stem cells for the treatment of complex perianal fistula including Crohn's disease. Expert Opin Biol Ther. 2008 Sep;8(9):1417-23. doi: 10.1517/14712598.8.9.1417. PMID 18694359
- [Derived] Garcia-Arranz M, Herreros MD, Gonzalez-Gomez C, de la Quintana P, Guadalajara H, Georgiev-Hristov T, Trebol J, Garcia-Olmo D. Treatment of Crohn's-Related Rectovaginal Fistula With Allogeneic Expanded-Adipose Derived Stem Cells: A Phase I-IIa Clinical Trial. Stem Cells Transl Med. 2016 Nov;5(11):1441-1446. doi: 10.5966/sctm.2015-0356. Epub 2016 Jul 13. PMID 27412883